CLINICAL TRIAL: NCT04793048
Title: A Randomized, Double-blind, Controlled Study to Evaluate the Safety and Feasibility of a Noninvasive Intraoral Electrotherapy Device for the Treatment of Patients With Periodontitis
Brief Title: A Randomized, Double-blind, Controlled Study to Evaluate the Safety and Feasibility of a Intraoral Electrotherapy Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Keku Medical Technology Co., Ltd. (Industry)
Collaborators: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91310110MA1G89RL54
Record Dates: First submitted 2021-03-10; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Root Planing

STUDY DESIGN:
Intervention Model Description: This trial was a parallel-arm, sham-controlled, randomized, and double-blind pivotal trial. A total of 30 patients were randomly assigned to one of two groups: one group received an active intraoral electrotherapy device and a scaling and root planing (SRP) at baseline, another group received a sham device and a scaling and root planing (SRP) at baseline.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Maintenance of blinding in this study was facilitated by the fact that (1) treatment delivery (active or sham) was hard-coded into the device's firmware, making active devices physically indistinguishable from sham devices, (2) both the device serial code block sizes and the treatment allocation block sizes were not known by the clinical investigative staff and that the order of blocks in each sequence was random, (3) patients only received treatment with their assigned device (active or sham) at home and never came in contact with another enrolled patient or device other than their own. This scheme rendered deliberate and accidental "breaking of the blind" difficult for both the patients or the clinical investigator, as no comparisons could be made between two devices that delivered different treatments and no pattern linking the device serial code and assigned treatment could be deduced, since the size and the order of blocks were randomly shuffled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group received an active device and a scaling and root planing (SRP) at baseline (Active Comparator)
  Interventions: Device: a noninvasive intraoral electrotherapy device
- Sham group received a sham device and a scaling and root planing (SRP) at baseline (Sham Comparator)
  Interventions: Device: a sham device

INTERVENTIONS:
Device: a noninvasive intraoral electrotherapy device — a noninvasive intraoral electrotherapy device to treat periodontal disease at-home for 20 minutes a day
  Other Names: a scaling and root planing (SRP)
  Arms: Active group received an active device and a scaling and root planing (SRP) at baseline
Device: a sham device — a sham device to be used at-home for 20 minutes a day
  Other Names: a scaling and root planing (SRP)
  Arms: Sham group received a sham device and a scaling and root planing (SRP) at baseline

SUMMARY:
A parallel-armed, sham-controlled, and participant-blind pilot study will be conducted to determine the safety and effectiveness of use of a noninvasive intraoral electrotherapy device to treat periodontal disease. A total of 30 patients were randomly assigned to one of two groups. The trial was comprised of three in-office oral examinations, which were performed at baseline, and at follow-ups～6 weeks (42 days ± 3 days) and～3months (84 days ± 3 days later).

DETAILED DESCRIPTION:
A parallel-armed, sham-controlled, and participant-blind pilot study will be conducted to determine the safety and effectiveness of use of a noninvasive intraoral electrotherapy device to treat periodontal disease at-home for 20 minutes a day. A total of 30 patients were randomly assigned to one of two groups: one group received an active intraoral electrotherapy device and a scaling and root planing (SRP) at baseline, another group received a sham device and a scaling and root planing (SRP) at baseline. The trial was comprised of three in-office oral examinations, which were performed at baseline, and at follow-ups～6 weeks (42 days ± 3 days) and～3months (84 days ± 3 days later). After 3 months of treatment, the effectiveness of the intraoral electrotherapy device would be demonstrated by (1) statistically superior reductions in the probing depth and clinical attachment level compared to treatment with the sham device. (2) statistically superior reductions in the bleeding on probing and gingival index compared to treatment with the sham device.

ELIGIBILITY:
Inclusion Criteria

1. Periodontitis at Stage Ⅲ having:

   i. Interdental CAL at site of greatest loss ≥5mm ii. Radiographic bone loss extending to mid-third of root and beyond iii. Tooth loss due to periodontitis ≤4 teeth IV. PD ≥ 6mm V. ≥30% of teeth involved
2. Participant has not had any treatment of periodontal disease in the six months
3. Participant is between the ages of 18 and 65 years inclusive.
4. Participant has read, signed and received a copy of the Informed Consent and HIPAA authorization prior to study initiation.
5. Participant is able to follow verbal and/or written instructions, perform oral hygiene procedures and return to the test facility for specified study examinations.

Exclusion Criteria

1. Participant has an implanted electrical stimulation device, such as a cardiac pacemaker, cardiac defibrillator, or deep brain stimulator.
2. Participant with oral cancer or oral mucosal diseases, or oral wound
3. Participant has any of the following:

   i. Fixed orthodontic appliances; or ii. Any metallic or amalgam crowns and/or restorations that have exposed metallic or amalgam surfaces at the gingival margin on both the buccal and lingual surfaces that, based on the clinical examiner's judgement, would inhibit proper function of the mouthpiece.
4. Participant has disqualifying acute or chronic medical illness as judged by the Principal Investigator.
5. Patients with specific allergic constitution, such as silica gel goods allergy
6. Participant is a smoker
7. Participant is pregnant or plans to become pregnant
8. Participant who have received other clinical research drugs or treatments within 3 months
9. The researchers considered that the subjects were not suitable for the clinical study because of other serious systemic diseases or other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-22 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Reductions in the probing depth | 3 months
Reductions in the clinical attachment level | 3 months

SECONDARY OUTCOMES:
Reductions in the bleeding on probing and gingival index | 3 months

IPD SHARING:
Plan to Share IPD: No